CLINICAL TRIAL: NCT04190784
Title: Optimal Duration of Stretching Exercises for Chronic Non-specific Neck Pain Patients:Randomized Controlled Trial
Brief Title: Optimal Duration of Stretching Exercises for Chronic Non-specific Neck Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Ibrahim Moustafa, Associate professor-chair of Physiotherapy Department, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Sharjah
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Myofascial Pain Syndrome
Keywords: Randomized controlled trial; Myofascial Pain Syndrome; Stretching exercises; nerve root function
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: A prospective, double blinded, parallel-group, randomized clinical trial was conducted at one of our university's research departments,
Who Masked: Participant, Investigator
Masking Description: The treating therapist, for both the control and intervention groups, was unblinded to the treatment method but the subjects and assessor who conducted the measurements were blinded. Assessor blinding was obtained through an independent research assist; not knowing the study design and not specifically involved in any aspect of the trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 60 seconds stretching group (Experimental): Stretching exercises for upper Trapezius and Levator scapula .
  From supine position , the examiner will passively place the participant's head into flexion, side-bending away and rotation towards the side to be stretched (for upper trapezius muscle) and flexion, side-bending away and rotation away from the side to be stretched (for levator scapula ). The patient introduces a light resisted effort to take the stabilized shoulder towards the ear and the ear towards the shoulder. The contraction is sustained for 10 seconds and, upon complete relaxation of effort, the therapist gently eases the head/ neck into an increased degree of side-bending and rotation, where it is stabilized, as the shoulder is stretched caudally. The examiner will depress the participant's shoulder with 100 Newton's of force measured with pressure dynamometer. Once the examiner achieved this level of force, he maintains the stretch for 60 seconds . The procedure is repeated three times.
  Interventions: Other: Stretching exercises
- 30 seconds stretching group (Experimental): The same procedures while the therapist will maintain the stretch for 30 seconds.
  Interventions: Other: Stretching exercises
- 15 seconds stretching group (Experimental): The same procedures while the therapist will maintain the stretch for 15 seconds.
  Interventions: Other: Stretching exercises
- 60 seconds placebo stretching group (Placebo Comparator): The therapist will maintain the same manual contact without stretching force for 60 seconds
  Interventions: Other: Placebo stretching
- 30 seconds placebo stretching group (Placebo Comparator): The therapist will maintain the same manual contact without stretching force for 30 seconds
  Interventions: Other: Placebo stretching
- 15 seconds placebo stretching group (Placebo Comparator): The therapist will maintain the same manual contact without stretching force for 15 seconds
  Interventions: Other: Placebo stretching

INTERVENTIONS:
Other: Stretching exercises — Post-facilitation stretch is a technique involves a maximal contraction of the muscle at mid-range with a rapid movement to maximal length followed by a static stretch.
  Other Names: Janda's post facilitation stretch method
  Arms: 15 seconds stretching group; 30 seconds stretching group; 60 seconds stretching group
Other: Placebo stretching — The therapist maintains the same manual contact without stretching force.
  Arms: 15 seconds placebo stretching group; 30 seconds placebo stretching group; 60 seconds placebo stretching group

SUMMARY:
A multitude of stretching parameters are used in the clinical setting. However, there is no convincing evidence to suggest which parameters are most effective in the management of chronic myofascial pain syndrome .In this regard, although the stretching duration is considered one of the most important variables that can affect the treatment outcome, to date there is little agreement on the most effective stretching duration.Accordingly ,we will conduct this study to investigate the effect of different stretching duration on nerve root function ,central conduction time, and chronic myofascial pain management outcomes.

DETAILED DESCRIPTION:
As Upper trapezius and levator scapulae are the most common postural muscles that tends to get shorten leading to restricted neck mobility as they are most frequently used to maintain posture,there seems to be strong rationale for stretching these muscles however, to date there is no agreement about the optimal stretching parameters . A multitude of stretching parameters are used in the clinical setting. However, there is no convincing evidence to suggest which parameters are most effective in the management of Chronic myofascial pain syndrome . In this regard, although the stretching duration is considered one of the most important variables that can affect the treatment outcome, to date there is little agreement on the most effective stretching duration.

In theory, reflex inhibition during the stretching procedure, an increased stretch tolerance , decreased viscoelasticity, and a degree of reduced musculotendinous stiffness could all contribute to the sustained increase in elastic ROM. Regardless of these proven underlying mechanisms, all the previous studies ignored the adverse mechanical tension that developed during stretching exercises . Based on the literature, this tension may adversely affect the central nervous system and nerve root function . Accordingly, in the current study ,we will try to answer the question that is it theoretically possible, that increased longitudinal stress and strain on the spinal cord and nerve root from stretching exercises may subtly impair the neural function.in addition to investigate the effect of stretching on other management outcomes;pain intensity,disability,range of motion,and Pressure-pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients will be included if they have active, palpable Myofascial trigger points on a single side or both sides of the upper trapezius muscle. Diagnosis was made according to Simons criteria, which includes five major and three minor criteria. For inclusion, cervical myofascial pain syndrome will be diagnosed with all five major criteria and at least one minor criterion.

Major criteria:

1. Regional pain complaint in the neck.
2. Pain complaint or altered sensation in the expected distribution of referred pain from a myofascial trigger point.
3. Taut band palpable in an accessible muscle.
4. Excruciating spot tenderness at one point along the length of the taut band.
5. Some degree of restricted range of motion , when measurable.

Minor criteria:

1. Reproduction of clinical pain complaint, or altered sensation, by pressure on the tender spot.
2. Elicitation of a local twitch response by transverse snapping palpation at the tender spot or by needle insertion into the tender spot in the taut band.
3. Pain alleviated by elongating (stretching) the muscle or by injecting the tender spot (trigger point).

Exclusion Criteria:

Participants will be excluded if any signs or symptoms of medical "red flags" were present: tumor, fracture, rheumatoid arthritis, osteoporosis, and prolonged steroid use. Additionally, subjects will be excluded with previous spine surgery and any exam findings consistent with neurological diseases and vascular disorders.

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
The change in peak-to-peak amplitudes of dermatomal somatosensory evoked potentials for C4,C5,C6,C7,&C8 | will be measured at two intervals ;pre-treatment and immediately after treatment
  Dermatomal Somatosensory Evoked Potentials will be elicited by repetitive, square wave (0.5 ms) electrical pulses (at 3 Hz) from standard clinical surface gel electrodes (20 mm) overlying cervical sensory dermatomes. Dermatomal somatosensory evoked potential will be collected at a stimulus intensity well above perception threshold.Complete recording runs will be undertaken during each session with averages of 250 to 1200 cortical responses from scalp surface recording electrodes (C3'-C4' in a 10-20 electrode configuration) of the contralateral scalp to the C4 to C8 dermatomes being stimulated

SECONDARY OUTCOMES:
The change in central conduction time | will be measured at two intervals ;pre-treatment and immediately after treatment.
  For central somatosensory conduction time measurement, N13-N20 will be determined for each subject following standard clinical procedure for upper limb stimulation (median nerve at the wrist). The difference in peak latency between N13 and N20 will be measured as central conduction time.
The change in Neck Disability Index | will be measured at two intervals ;pre-treatment and immediately after treatment.
  The Neck Disability Index , consisting of 10 items related to daily living activities, will be our primary patient-reported outcome measure.
The change in Cervical range of motion | will be measured at two intervals ;pre-treatment and immediately after treatment
  Cervical spine global range-of-motion will be measured using the valid and reliable cervical range-of-motion (CROM) device. The participant will perform flexion, extension, right/left lateral flexion, right/left rotation in upright sitting. The patient was instructed to perform each movement when he/she attained the maximum active range of motion. Three trials were conducted for each direction of movement, and the average of the three measurements will be recorded for analysis.
The change in Neck pain intensity | will be measured at two intervals ;pre-treatment and immediately after treatment
  Neck pain intensity will be measured using the numerical pain rating scale . The patients will be asked to place a mark along the line indicating their current pain intensity; 0 reflecting ''no pain'' and 10 reflecting the ''worst pain''.
The change in Pressure-pain threshold , algometric measurement | will be measured at two intervals ;pre-treatment and immediately after treatment.
  A pressure threshold algometer will be used to measure pressure-pain threshold in the most tender point of the upper trapezius and levator muscles. The average value of 3 repetitive measurements with an interval of 30 to 60 seconds will be taken for data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M Moustafa, Assoc prof, Study Director — University of Sharjah
Locations (1):
- Ibrahim Moustafa, Sharjah city, United Arab Emirate, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data and related data dictionaries available
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months and will become available for one year
Access Criteria: not identified yet

REFERENCES:
- [Background] Backes WH, Nijenhuis RJ (2008): Advances in spinal cord MR angiography. AJNR Am J Neuroradiol ; 29(4):619-31. Biglioli, Paolo; et alia (2004): Upper and lower spinal cord blood supply: the continuity of the anterior spinal artery and the relevance of the lumbar arteries. Journal of Thoracic and Cardiovascular Surgery 127 (4): 1188-1192. Challis, J.H. (1995): A procedure for determining rigid body transformation parameters. J Biomech 28, 733-737. Cheung, Karoline, Patria A. Hume, and Linda Maxwell. (2003): Delayed Onset Muscle Soreness: Treatment Strategies and Performance Factors.